CLINICAL TRIAL: NCT05764720
Title: A Prospective Trial of Stereotactic Adaptive Radiation Therapy for Borderline Resectable/Locally Advanced Pancreatic Cancer: An Individualized Approach to Minimizing Gastrointestinal Toxicity (ARTIA-Pancreas)
Brief Title: Stereotactic Adaptive Radiation Therapy of Borderline Resectable Pancreatic Cancer an Individualized Approach
Acronym: ARTIA-Pancreas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-07
Record Dates: First submitted 2023-02-13; First posted 2023-03-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Daily Adaptive External Beam Radiation Therapy (Experimental): Daily adaptive radiation therapy delivered with Varian Ethos treatment system
  Interventions: Radiation: Daily Adaptive External Beam Radiation Therapy

INTERVENTIONS:
Radiation: Daily Adaptive External Beam Radiation Therapy — Daily adaptive external beam radiation therapy delivered on Varian Ethos treatment system.

SUMMARY:
This trial is a single-arm, prospective, multi-center clinical trial designed to demonstrate that stereotactic adaptive radiotherapy using an ablatively dosed (50Gy,5fx) for treatment of borderline-resectable, locally-advanced , or medically inoperable pancreatic adenocarcinoma will translate into a decreased toxicity. The study will evaluate GI toxicity, overall survival, local control, quality of life, and workflow metrics.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed borderline-resectable (based on NCCN criteria), locally-advanced (based on NCCN criteria), or medically inoperable pancreatic adenocarcinoma.
2. ECOG performance status 0-1
3. Receipt of at least two months of lead-in chemotherapy (regimen at the discretion of the treating physician) prior to planned initiation of CT-STAR.
4. Limited regional lymphadenopathy permitted. Node positive patients are restricted to those with up to 3 clinically involved (greater than 1cm on cross-sectional imaging or pathologically proven) nodes provided that the lymph nodes are adjacent to the primary tumor.
5. At least 18 years of age.
6. Must be able to take an interruption in systemic therapy at least one week prior to planned start of CT-STAR (two weeks preferred) lasting for the duration of CT-STAR and continuing for at least one week following end of CT-STAR (two weeks preferred).
7. Capable of a single end-exhale breath-hold of at least 20 seconds in duration and of repeated end-exhale or deep inspiratory breath-hold of at least 10 seconds in duration upon verbal instruction.
8. Anatomy of target and adjacent OARs adequately visualized on ETHOS simulation imaging, as determined by treating and study physicians.

   Note: central review of simulation imaging and initial plan target/OAR contours by the Principal Investigator and Physics lead is required for the first two patients at each participating institution prior to study treatment delivery. Patients with inadequate anatomic visualization at simulation will be considered screen-failures and treated off-protocol as per institutional standard-of-care.
9. Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

1. Past history of radiotherapy within the projected treatment field
2. Prior, intercurrent, or planned receipt (within 90 days prior to or following SBRT) of any investigational agents related to pancreatic cancer diagnosis.
3. Competing, active cancer diagnosis within the preceding one year.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Gross tumor invasion of the stomach or duodenum (defined either radiographically or endoscopically).
6. Pregnant and/or breastfeeding. Patients of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-05-14 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Acute Grade 3+ treatment related GI toxicities | Within 90 days from start of treatment
  The rate of acute Grade 3 or higher treatment related GI toxicities using CTCAE version 5.0 criteria

SECONDARY OUTCOMES:
Long Term Grade 3+ treatment related GI toxicities | 12 months after completion of external beam radiation treatment
  The rate of long term Grade 3 or higher treatment related GI toxicities, using CTCAE version 5.0 criteria
Overall Survival | One and two years after completion of external beam radiation treatment
  Kaplan-Meier estimates of the rates of overall survival
Local in-field Control | One and two years after completion of external beam radiation treatment
  Local (in-field) control rates defined as stable disease, partial response, or complete response by RECIST criteria
Progression Free Survival | One and two years after completion of external beam radiation treatment
  Kaplan-Meier estimates of distant-progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Henke, MD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Washington University, St. Louis, St Louis, Missouri
  - UH Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No